CLINICAL TRIAL: NCT02901717
Title: Efficacy and Safety of Mino-Lok Therapy (MLT) in Combination With Systemic Antibiotics in the Treatment of Catheter-Related or Central Line-Associated Bloodstream Infection
Brief Title: Mino-Lok Therapy (MLT) for the Treatment of CRBSI/CLABSI
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leonard-Meron Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MDA-2013-0039
Record Dates: First submitted 2016-08-31; First posted 2016-09-15 (Estimated); Last update posted 2022-04-19 (Actual); Status verified 2021-07

CONDITIONS: Catheter-related Infections
MeSH Terms: conditions — Catheter-Related Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): Antibiotic lock + standard of care antibiotics. The standard of care antibiotic will be chosen by the investigator at the time of the infection.
  Interventions: Drug: Antibiotic lock
- Mino-Lok Therapy (MLT) (Experimental): Standard of care plus MLT. MLT contains minocycline with EDTA and ethanol.
  Interventions: Drug: Mino-Lok

INTERVENTIONS:
Drug: Mino-Lok — Standard of Care antibiotics appropriate for the infecting organism plus Mino-Lok therapy to disinfect and save the catheter.
  Other Names: Standard of care antibiotics + Mino-Lok
  Arms: Mino-Lok Therapy (MLT)
Drug: Antibiotic lock — Standard of Care antibiotics appropriate for the infecting organism with an antibiotic lock solution using the same standard of care antibiotic delivered systemically. The antibiotic lock arm may include subjects with S. aureus, including methicillin-resistant S. aureus, vancomycin intermediate S. aureus, or vancomycin-resistant S. aureus; vancomycin resistant enterococci; Candida, Pseudomonas; other Gram negative organisms; or other organisms deemed to be of high virulence per the Investigator. The standard of care antibiotic will be determined by the investigator at the start of treatment.
  Other Names: Standard of Care antibiotics with antibiotic lock
  Arms: Standard of Care

SUMMARY:
This is a Phase 3, multi-center, randomized, open-label, assess-blind study to determine the efficacy and safety of MLT, a novel antibiotic lock therapy that combines minocycline with edetate disodium in 25% ethanol solution as an adjuctive therapy for the treatment of catheter-related or central line associated bloodstream infection (CRBSI/CLABSI).

Approximately 144 subjects who have been diagnosed with CRBSI/CLABSI and who meet all necessary criteria for the study will be randomized in a 1:1 ratio to 1 of 2 treatment arms:

* MLT Arm: Mino-Lok therapy; or
* Control Arm: Antibiotic lock (±heparin). The antibiotic lock (ALT) should be comprised of the best available therapy at the sites based on standard institutional practices or recommendations from the Infectious Diseases Society of America (IDSA) guidelines.

DETAILED DESCRIPTION:
This is a Phase 3, multi-center, randomized, double-blind study to determine the efficacy and safety of MLT, a novel antibiotic lock therapy that combines minocycline with edetate disodium in 25% ethanol solution.

Mino-Lok Therapy is being developed as an adjunctive therapy for the treatment of catheter-related or central line associated bloodstream infection (CRBSI/CLABSI) in combination with appropriate systemic antibiotic(s), to preserve central venous access and to avoid the complications and morbidities associated with catheter removal and reinsertion.

Approximately 144 subjects who have been diagnosed with CRBSI/CLABSI and who meet all necessary criteria for the study will be randomized in a 1:1 ratio to 1 of 2 treatment arms:

* MLT Arm: MLT + SOC intravenous (IV) antibiotic therapy; or
* Control Arm (subjects randomized to the Control Arm will receive treatment based on the type and virulence of the infecting organism as documented by the Investigator prior to randomization): The antibiotic lock should be comprised of the best available therapy at the sites. Prior to randomization, the Investigator at each site will determine the antibiotic used in the lock, the dose, the dwell time, and the number of days of administration (minimum of 7 days) based on standard institutional practices or recommendations from the Infectious Diseases Society of America (IDSA) guidelines. In the event that the subject is being treated with more than 1 systemic SOC IV antibiotic, the Investigator will specify a single antibiotic that should be used for the antibiotic lock. It is acceptable for the SOC antibiotic lock to differ from the SOC IV antibiotics, as necessary per local SOC.

All infecting organism types are permitted (eg, S. aureus, S. epidermidis, Candida spp., Pseudomonas aeruginosa). Randomization will be stratified by type of CVC, presence of neutropenia, and by virulence of the infecting organism.

The primary endpoint for this study is the time (in days following randomization) to a catheter failure event between randomization and TOC (Week 6) in the Intent-to-Treat (ITT) Population.

A catheter failure event is ANY of the following:

* All-cause mortality at TOC (Week 6). The event time is the day of death;
* Catheter removal for any infection-related reasons (including worsening of symptoms or failure to eradicate the infection). The event time is the day the catheter is removed;
* Inability to administer study drug. The event time is the day the Investigator determines the catheter is no longer functional;
* Worsening of systemic signs and symptoms of infection that result in change in systemic anti infective treatment. Note that changes in treatment based on susceptibility data will be permitted. The event time is the day the treatment is changed;
* Demonstration that the baseline pathogen is not eradicated from the blood culture collected within 72 hours following randomization despite 72 hours of antibiotic therapy to which the infecting organism is susceptible. Best clinical practice and subject safety may dictate changes in treatment prior to 72 hours. The event time is the day of the positive culture;
* Demonstration that the baseline pathogen has recurred based on blood culture results by Week 6 of the study. The event time is the day of the positive blood culture documenting the recurrence. If a subject does not show any signs and symptoms of an infection and there is a negative blood culture prior to Week 6, then a blood culture does not have to be performed at Week 6. Subjects whose catheter was removed for reasons not related to the baseline infection also do not need to have a blood culture at Week 6; or
* Demonstration that the baseline pathogen is part of a newly diagnosed deep-seated infection by Week 6 of the study. The event time is the day of the new diagnosis.

Removal of the CVC prior to TOC because the catheter is no longer needed will not be considered a catheter failure and these subjects will be censored at the time of catheter removal.

ELIGIBILITY:
Subjects with CRBSI/CLABSI for whom, in the Investigator's opinion, catheter retention is reasonable or required due to lack of alternative venous access. This includes subjects with bacterial pathogens and Candida spp.

Inclusion Criteria

1. Subject or a legally authorized representative must provide a signed informed consent form;
2. Male or female at least 12 years of age;
3. Subject must have a bloodstream infection with no other apparent source other than the CVC that meets one of the following criteria:

   * A recognized single pathogen cultured from 1 or more blood cultures; OR
   * A common skin contaminant cultured from 2 or more blood cultures drawn on the same or consecutive calendar days from a subject with fever (greater than or equal to 38.0 degrees C), chills, or hypotension (systolic blood pressure less than 90 mmHg); NOTE: When possible, it is recommended to collect from both the CVC and peripheral venipuncture.
4. Inpatient or outpatient with presence of indwelling CVC (ie, totally implantable port, tunneled or non-tunneled CVC, hemodialysis catheter, or peripherally inserted CVC) that has been in place for at least 5 days;
5. A bloodstream infection documented within 96 hours prior to enrollment (and from which an isolate of the baseline pathogen(s) is still available for analysis at the central laboratory) and demonstrates the protocol definition of CRBSI or CLABSI;

   NOTE: Subjects may be enrolled and randomized while awaiting results of standard blood cultures from the local laboratory:
   * If an organism has been identified from blood specimen testing using an FDA-cleared rapid diagnostic test (eg, T2MR®); or
   * If a positive blood culture specimen shows an organism by 1 of the following:

   Gram stain; or An FDA-cleared molecular rapid diagnostic test (eg, FilmArray® BCID or Verigene®); If the pending blood culture does not confirm a qualifying organism by standard methods and an isolate is not available for testing at the central laboratory, the subject will be withdrawn from study drug treatment and managed at the Investigator's discretion.

   NOTE: Subjects with a positive blood culture identified up to 120 hours prior to enrollment and in whom the baseline pathogen is still available for analysis at the central laboratory may be considered on a case by-case basis with prior approval from the Medical Monitor.
6. Subjects for whom, in the Investigator's opinion, catheter retention for the duration of the study (6 weeks) is reasonable or required;
7. Female subjects of childbearing potential must have a negative urine and/or serum pregnancy test within 5 days prior to randomization;

   NOTE: The following are considered women who are NOT of childbearing potential:
   * Postmenopausal (defined as no menses for at least 12 consecutive months); or
   * Documented to be surgically sterile;
8. Female subjects of childbearing potential and male subjects who are sexually active must agree to use a highly effective method of contraception from the time of informed consent until 30 days post dose; NOTE: Highly effective methods of contraception include hormonal contraceptives, intrauterine device, double-barrier method, partner sterility, or abstinence.
9. Male subjects must agree to refrain from sperm donation throughout the duration of the study and for 90 days following the last dose of study drug; and
10. Subject must be willing to comply with all study procedures, whether inpatient or outpatient, for the duration of the study.

Exclusion Criteria

1. Subjects with hypersensitivity or allergy to tetracycline antibiotics or edetate disodium;
2. Subjects with septic shock that requires inotropic support or is unresponsive to fluid resuscitation;
3. Subjects taking disulfiram at the time of randomization or who are expected to take disulfiram at any time during treatment with study drug;
4. Subjects with prosthetic cardiac valves, vascular grafts, pacers, automatic implantable cardioverter-defibrillator, or other non-removable vascular foreign body, with the exception of coronary stents and peripheral stents;
5. Subjects with the presence of a deep-seated intravascular source of infection (eg, endocarditis [as evidenced by vegetations on an echocardiogram or clinical suspicion] or septic thrombosis);
6. Subjects with bacteremia with documented microbiological evidence of another source of infection (eg, osteomyelitis, pneumonia, skin infection, urinary tract infection, joint infection, or abdominal infection) known to be due to the same organism cultured from the blood;
7. Subjects with polymicrobial CRBSI/CLABSI caused by pathogens that would require multiple antibiotics to be used for adequate lock therapy treatment. For example, a subject with methicillin-resistant Staphylococcus aureus and Escherichia coli requiring treatment with vancomycin and meropenem would be excluded from the study. A subject with S. aureus and Staphylococcus epidermidis, where both are identified as pathogens and where both could be treated with vancomycin, would be eligible; NOTE: If more than 1 organism is isolated, the Investigator should decide which of the organisms are pathogens and require therapy. Isolates of all organisms should be sent to the central laboratory. In the event that the subject is being treated with more than 1 systemic standard of care (SOC) anti-infective, the Investigator will specify a single antibiotic that should be used for the antibiotic lock. It is acceptable for the SOC antibiotic lock to differ from the SOC anti infectives, as necessary per local SOC.
8. Subjects with the presence of a tunnel or catheter exit site infection or an infusion port pocket abscess as manifested by purulence at the exit site, or inflammation with erythema, or induration of at least 1 cm in diameter;
9. Subjects who have been previously randomized into the present study;
10. Subjects who are pregnant or breastfeeding;
11. Subjects with proven or suspected persistent bacteremia or fungemia despite 72 hours of both systemic anti-infective therapy and lock therapy to which the infecting organism is susceptible;
12. Subjects with short-term CVCs indwelling at least 5 days;
13. Subjects with a central line-related mycobacterial infection or fungi other than Candida; or
14. Subjects who, in the opinion of the Investigator, have a high probability of death within 3 months of randomization due to a disease process other than the CRBSI/CLABSI.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2018-02-13 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Time to a catheter failure event. | 6 weeks
  The time (in days following randomization) to a catheter failure event between randomization and TOC (Week 6) in the Intent-to-Treat (ITT) Population.

SECONDARY OUTCOMES:
Proportion of subjects with overall success in the MITT and CE populations. | 6 weeks
  Overall success is defined as no catheter failure events by TOC (week 6).
Time to catheter failure in the MITT and CE Populations. | 6 weeks
  The time (in days following randomization) to a catheter failure event between randomization and TOC (Week 6).
Microbiological eradication | 6 weeks
  Proportion of subjects with Microbiological Eradication at TOC (Week 6) in the MITT and CE Populations.
Clinical Cure | 6 Weeks
  Proportion of subjects with Clinical Cure at TOC (Week 6) in the MITT and CE Populations.
  Clinical Cure is defined as the absence of baseline CRBSI/CLABSI signs/symptoms or, in the Investigator's opinion, improvement of signs/symptoms such that no additional therapy is necessary.
All-cause mortality | 6 weeks
  Death within 6 weeks of randomization
Safety and Tolorability | 6 Weeks
  Safety and tolerability profile as assessed by adverse events, serious adverse events (SAEs), vital signs, clinical laboratory evaluations, and physical examinations.

CONTACTS AND LOCATIONS:
Locations (22):
- United States (19):
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Florida Shands Hospital, Gainesville, Florida
  - Edward Hines Jr. VA Hospital, Hines, Illinois
  - AMG Oncology, Park Ridge, Illinois
  - Indiana Blood and Marrow Institute, Indianapolis, Indiana
  - Ascension Via Christi Hospital, Wichita, Kansas
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Anne Arundel Medical Center, Annapolis, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Health Systems, Detroit, Michigan
  - William Beaumont Hospital, Troy, Michigan
  - VA Sierra Nevada Health Care Systems, Reno, Nevada
  - Saint Michael's Medical Center, Newark, New Jersey
  - Carolinas Medical Center, Charlotte, North Carolina
  - East Carolina University, Greenville, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Salem VA Medical Center, Salem, Virginia
  - Seattle Children's Hospital, Seattle, Washington
- Puerto Rico (3):
  - VA Caribbean Healthcare System, San Juan, PR
  - Manati Medical Center, Manatí
  - Ponce Research Institute, Ponce

IPD SHARING:
Plan to Share IPD: No